CLINICAL TRIAL: NCT06264986
Title: The Effects of Ashwagandha (Withania Somnifera) Supplementation on Exercise Performance in Female Footballers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blanca Roman-Viñas, MD (Other)
Responsible Party: Sponsor-Investigator, Blanca Roman-Viñas, MD, Professor, University Ramon Llull
Organization: University Ramon Llull (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023-09-02
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Muscle Strength
MeSH Terms: interventions — Ashwagandha

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomised trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KSM-66 (Experimental): 600mg (5% withanolides) KSM-66 ashwagandha, hydroxypropyl methylcellulose capsule
  Interventions: Dietary Supplement: Ashwagandha
- Placebo (Placebo Comparator): 600mg Gluten-free chickpea powder, hydroxypropyl methylcellulose capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ashwagandha — The intervention will be 600mg of KSM-66, a branded supplement derived from the root extract of the herb ashwagandha, with a consistent rate of 5% withanolides for 28 days. It is the most clinically studied extract of the herb and is the only type of ashwagandha to receive third party testing certification (Informed Sport, Informed Ingredient, Banned Substances Control Group, Clean Label Project). The laboratory where the product is made, Ixoreal Biomed, has received Current Good Laboratory Practices (cGLP), quality controlled and tested against heavy metals and pesticides.
  Other Names: KSM-66; Root extract ashwagandha
  Arms: KSM-66
Other: Placebo — 600mg chickpea flour in a hydroxypropyl methylcellulose capsule, once a day for 28 days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effects of short-term root extract ashwagandha supplementation on exercise performance in female footballers. The main question it aims to answer are:

Will short-term supplementation of root extract ashwagandha improve muscle strength markers in female footballers? Will short-term supplementation of root extract ashwagandha improve perception of recovery following high-intensity exercise in female footballers?

Participants will either supplement 600mg (5% withanolides) root extract ashwagandha or placebo once a day for 28 days. There will be three data points: baseline, 14 days and 28 days. Researchers will compare values of intervention against placebo to see if there is an effect on muscle strength or perception of recovery.

DETAILED DESCRIPTION:
The objectives of the thesis are to determine the effects of ashwagandha (ASH) on muscle strength, muscle recovery and to assess habitual dietary intake of female footballers. Across one phase, two experimental research papers and one descriptive research paper will be produced; it will involve one double-blind, randomised and placebo-controlled trial and a comparative analysis of nutritional intake in female footballers. The thesis will involve participants supplementing ASH in the form of a capsule containing KSM-66 (600 mg with 30mg withanolides) or placebo once a day for 28 days, on a singular occasion. The objectives of the first two papers are to determine the effects of ASH on muscle strength, perception of recovery, perception of exertion, perceived wellness and perceived muscle soreness. For the paper on muscle strength, the methodology will include hand grip test, counter movement jump (CMJ), squat jump (SJ), peak power, medicine ball throw and rate of perceived exertion (RPE) via the Borg Scale. For the paper on muscle recovery, the methodology will include a questionnaire on sleep, stress, fatigue and delayed onset of muscle soreness (DOMS) test via the Hooper Index (HI), total quality recovery (TQR) questionnaire and a supplement satisfaction questionnaire. The objectives of the third paper are to evaluate the dietary intake of professional female footballers and compare the values against published nutritional recommendations. The participants diets will be tracked for purposes of the muscle strength and recovery study. The methodology will involve self-tracking of dietary intake via the Snap-N-Send method and data will be stored and analysed with the software Nutritics. The study will be conducted with a professional club in Barcelona. The use of ASH is becoming prevalent in athletes, despite lack of information regarding dosage guidelines or lack of research on its benefits for exercise performance. The proposed study will contribute to the overall scientific knowledge of ASH and whether it may demonstrate benefits from short-term use. Additionally, the study will determine if there are benefits for female athletes that wish to increase strength and reduce perception of pain or soreness related to exercise. The ethical considerations for this study are predominantly the safety and comfort of the participant. An informed consent form will be given to the participant, containing information about data collection, personal information, safety of the supplement and their right to drop out of the study at any point. The proposed start date is January 2024, and the study will aim to collectively last for 36 days across a singular phase. The supplement is provided by Zenement España, a supplement company based in Barcelona.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Playing football professionally
* At a sub-elite to elite standard
* Healthy and free of disease

Exclusion Criteria:

* Active supplementation with other ergogenic aids
* Medication or contraceptives (to not interfere with existing treatment)
* Thyroid conditions (due to interaction with cortisol)
* Diabetes or certain autoimmune conditions (to not interfere with existing treatment)
* Active pregnancy (to not interfere with existing treatment)
* Allergies to nightshades such as tomato, aubergine, potatoes and peppers
* No signing of the consent form

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants must be female or assigned female at birth
Enrollment: 30 (Actual)
Dates: Start 2024-01-13 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Roman Viñas, Principal Investigator — Blanquerna, Ramon Llull University
Locations (1):
- Club Esportiu Seagull, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonilla DA, Moreno Y, Gho C, Petro JL, Odriozola-Martinez A, Kreider RB. Effects of Ashwagandha (Withania somnifera) on Physical Performance: Systematic Review and Bayesian Meta-Analysis. J Funct Morphol Kinesiol. 2021 Feb 11;6(1):20. doi: 10.3390/jfmk6010020. PMID 33670194
- [Derived] Coope OC, Reales Salguero A, Spurr T, Paez Calvente A, Domenech Farre A, Jordan Fisas E, Lloyd B, Gooderick J, Abad Sangra M, Roman-Vinas B. Effects of Root Extract of Ashwagandha (Withania somnifera) on Perception of Recovery and Muscle Strength in Female Athletes. Eur J Sport Sci. 2025 Mar;25(3):e12265. doi: 10.1002/ejsc.12265. PMID 39954269

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KSM-66 | Placebo
Started | 15 | 15
Completed | 0 | 0
Not Completed | 15 | 15

BASELINE CHARACTERISTICS:
Population: Female, healthy, over 18 years of age, footballer assigned to a professional club.
Groups:
- Total: Total of all reporting groups
Arm/Group | KSM-66 | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Increased Lower Body Muscle Strength 1/2
Description: Jump strength, assessed by Peak Power, is calculated based on jump height (in centimetres) and body mass (in kilograms) using this formula Peak power (W) = (60.7) × (jump height [cm]) + 45.3 × (body mass [kg]) - 2055 [1]. Jumps are measured using a clinically validated open-source jump mat (Chronojump Bocosystems) to ensure accuracy. The highest recorded value is used for analysis.
  1. Sayers, S. P.; Harackiewicz, D. V.; Harman, E. A.; Frykman, P. N.; Rosenstein, M. T. Cross-Validation of Three Jump Power Equations. Medicine and science in sports and exercise 1999, 31 (4), 572-577. https://doi.org/10.1097/00005768-199904000-00013.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | KSM-66 | Placebo
Number analyzed (Participants) | 15 | 15
Watts | 2410.0 (82.5) | 2492.5 (96.6)

2. Primary Outcome: Increased Maximum Voluntary Muscle Strength
Description: Hand grip strength. This will be measured with a CAMRY digital hand dynamometer and the unit of measurement will be kilograms.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | KSM-66 | Placebo
Number analyzed (Participants) | 15 | 15
kilograms | 33.14 (1.5) | 31.8 (1.0)

3. Primary Outcome: Increased Upper Body Muscle Strength and Explosiveness
Description: Medicine ball throw using a 5 kilogram medicine ball. Participants will throw a medicine ball while standing. The distance of the throw will be measured in centimetres.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Centimetres
Arm/Group | KSM-66 | Placebo
Number analyzed (Participants) | 15 | 15
Centimetres | 160.7 (8.4) | 153.9 (7.9)

4. Primary Outcome: Improved Overall Muscle Strength
Description: Rate of perceived exertion (RPE) using the Borg Scale measuring the difficulty of high-intensity exercise. 1 represents a score of very light activity, and 10 represents a score of maximum effort activity.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | KSM-66 | Placebo
Number analyzed (Participants) | 15 | 15
Units on a scale | 6.1 (0.3) | 5.4 (0.5)

5. Secondary Outcome: Improved Perception of Wellbeing
Description: Hooper Index questionnaire. Participants rate their perception of sleep, stress, fatigue and muscle soreness on a scale. A score of 1 is very, very good and 10 is a score of very, very bad.
  The Hooper Index questionnaire assesses participants' perception of sleep quality, stress levels, fatigue, and muscle soreness. Each item is rated on a scale from 1 to 10, where 1 represents "very, very good" and 10 represents "very, very bad." The minimum possible score for each item is 1, and the maximum possible score is 10. Higher scores indicate a worse perception of wellbeing. An overall wellbeing score is calculated by summing scores for sleep, stress, fatigue, and muscle soreness, with a total range from 4 (very good) to 40 (very bad).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | KSM-66 | Placebo
Number analyzed (Participants) | 15 | 15
Units on a scale | 11.4 (1.2) | 13.5 (1.3)

6. Secondary Outcome: Improved Perception of Recovery
Description: Total Quality Recovery questionnaire. Participants rate their recovery following high-intensity exercise. A score of 6 is very, very low recovery and 20 is a score of very, very good recovery.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | KSM-66 | Placebo
Number analyzed (Participants) | 15 | 15
Units on a scale | 15.9 (0.6) | 14.0 (0.6)

7. Primary Outcome: Increased Lower Body Muscle Strength in 2/2
Description: Lower body muscle strength is assessed using the countermovement jump (CMJ) and squat jump (SJ) tests, two validated measures of lower body explosive power. Each participant performs a single jump for each test on a clinically validated open-source jump mat (Chronojump Bocosystems), which records jump height in centimetres. The jump mat uses precise force and time measurements to calculate height, ensuring reliable data output. Participants receive standardised instructions and a demonstration before testing to ensure consistency and accuracy.The highest recorded value is used for analysis.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Centimetres
Arm/Group | KSM-66 | Placebo
Number analyzed (Participants) | 15 | 15
Centimetres | 27.9 (1.0) | 28.7 (1.5)

ADVERSE EVENTS:
Time Frame: One month
Description: Adverse events were defined in accordance with ClinicalTrials.gov standards including any medical occurrences regardless of relation to the intervention. Serious adverse events included any events resulting in death, life-threatening situations, hospitalisation or significant disability. Data were collected over one month, with monitoring conducted weekly based on participant self-reports and investigator assessments. No differences in definition were applied from the standard ClinicalTrials.gov
Arm/Group | KSM-66 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
No clinical testing, such as blood biomarkers, to correlate physiological data with observed outcomes, limiting conclusions about ashwagandha's biochemical effects on muscle strength and recovery. Sleep quality was self-reported - future studies should use objective methods. The convenience sample limits generalisability, and larger samples are needed. Lack of a crossover design also restricts control over confounders, and future research could benefit from this approach to reduce variability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT06264986/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT06264986/ICF_001.pdf